CLINICAL TRIAL: NCT06731777
Title: Oral Gel Containing PHTALOX® as an Adjuvant in the Treatment of Periodontal Disease: A Randomized Controlled Clinical Trial
Brief Title: Oral Gel Containing PHTALOX® as an Adjuvant in the Treatment of Periodontal Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Alfenas (Other)
Responsible Party: Principal Investigator, Marcelo Franchin, Professor, Universidade Federal de Alfenas
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 39624820.6.0000.5142
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vehicle Group (Sham Comparator): Toothbrushing with dental gel and local application of the PHTALOX® oral gel vehicle
  Interventions: Procedure: Scaling and root planing plus PHTALOX® oral gel vehicle
- Chlorhexidine Group (Active Comparator): Toothbrushing with dental gel and local application of 0.12% chlorhexidine oral gel.
  Interventions: Procedure: Scaling and root planing plus 0.12% chlorhexidine oral gel
- PHTALOX® Group (Experimental): Toothbrushing with dental gel and local application of 1% PHTALOX® oral gel
  Interventions: Procedure: Scaling and root planing plus PHTALOX® oral gel

INTERVENTIONS:
Procedure: Scaling and root planing plus PHTALOX® oral gel vehicle — Root scaling and planing (RAR) will be performed following the full-mouth disinfection (FMD) protocol. After anesthesia using the regional block technique [2% lidocaine solution with 1:100,000 epinephrine (Nova DFL)], RAR will be conducted by an experienced professional using an ultrasonic scaler and periodontal curettes (Millenium Curettes, Golgran, São Paulo, Brazil). The time spent per quadrant will be approximately one hour. Polishing will then be performed using a rubber cup and prophylactic paste (Odahcam, Dentsply Sirona, USA). The oral gel (PHTALOX® oral gel vehicle) should be applied to all free dental surfaces using a plastic applicator with cotton tips. The contact between the gel and the tooth surface must last for 5 minutes. After this time, the patient should spit out the excess gel without rinsing the mouth. This process should be performed after the last brushing of the day for a period of 45 days.
  Arms: Vehicle Group
Procedure: Scaling and root planing plus 0.12% chlorhexidine oral gel — Root scaling and planing (RAR) will be performed following the full-mouth disinfection (FMD) protocol. After anesthesia using the regional block technique [2% lidocaine solution with 1:100,000 epinephrine (Nova DFL)], RAR will be conducted by an experienced professional using an ultrasonic scaler and periodontal curettes (Millenium Curettes, Golgran, São Paulo, Brazil). The time spent per quadrant will be approximately one hour. Polishing will then be performed using a rubber cup and prophylactic paste (Odahcam, Dentsply Sirona, USA). The oral gel (0.12% chlorhexidine oral gel) should be applied to all free dental surfaces using a plastic applicator with cotton tips. The contact between the gel and the tooth surface must last for 5 minutes. After this time, the patient should spit out the excess gel without rinsing the mouth. This process should be performed after the last brushing of the day for a period of 45 days.
  Arms: Chlorhexidine Group
Procedure: Scaling and root planing plus PHTALOX® oral gel — Root scaling and planing (RAR) will be performed following the full-mouth disinfection (FMD) protocol. After anesthesia using the regional block technique [2% lidocaine solution with 1:100,000 epinephrine (Nova DFL)], RAR will be conducted by an experienced professional using an ultrasonic scaler and periodontal curettes (Millenium Curettes, Golgran, São Paulo, Brazil). The time spent per quadrant will be approximately one hour. Polishing will then be performed using a rubber cup and prophylactic paste (Odahcam, Dentsply Sirona, USA). The oral gel (PHTALOX®) should be applied to all free dental surfaces using a plastic applicator with cotton tips. The contact between the gel and the tooth surface must last for 5 minutes. After this time, the patient should spit out the excess gel without rinsing the mouth. This process should be performed after the last brushing of the day for a period of 45 days.
  Arms: PHTALOX® Group

SUMMARY:
Periodontitis, a chronic inflammatory condition of the periodontal tissues, impacts not only the patient's oral and systemic health but also has significant social and economic implications. While mechanical treatment effectively removes calculus and dental biofilm, it may fail to eliminate pathogenic bacteria in soft tissues and in areas inaccessible to periodontal instruments, such as furcation regions, root concavities, interproximal areas, and deep periodontal pockets. Consequently, adjuvant therapies with antimicrobial and anti-inflammatory potential represent a valuable strategy for periodontitis treatment. In this context, an oral gel containing a phthalocyanine derivative, known for its antimicrobial and anti-inflammatory properties, offers a promising enhancement to conventional periodontal treatment. This randomized controlled clinical trial aimed to evaluate the effect of the topical application of an oral gel formulation containing iron tetracarboxyphthalocyanine (PHTALOX®) in the non-surgical periodontal treatment. Patients with periodontitis underwent a standard periodontal treatment protocol (scaling and root planing), followed by adjuvant therapy according to the assigned groups: Vehicle Group: Toothbrushing with dental gel and local application of the PHTALOX® oral gel vehicle. Chlorhexidine Group: Toothbrushing with dental gel and local application of 0.12% chlorhexidine oral gel. PHTALOX® Group: Toothbrushing with dental gel and local application of 1% PHTALOX® oral gel. Clinical evaluations (plaque index, probing depth, bleeding on probing, clinical attachment level, and mobility test) were performed at baseline (day 0) and post-treatment (day 45).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with periodontitis stages II to IV (moderate to severe) grades A-C, with at least two non-adjacent interproximal sites showing probing depth (PD) ≥5 mm, clinical attachment level (CAL) ≥3 mm, and bleeding on probing

Exclusion Criteria:

* Medical conditions requiring antibiotic prophylaxis or that could influence the response to treatment.
* History of periodontal treatment within the last 6 months.
* Use of medications affecting periodontal tissues within the last 3 months (antibiotics, anti-inflammatory drugs, anticonvulsants, immunosuppressants, or calcium channel blockers).
* Smokers or former smokers within the last 12 months.
* Pregnancy.
* Extensive prosthetic rehabilitation.
* Undergoing orthodontic treatment.
* Individuals with blood dyscrasias.
* Alcoholism.
* Use of illicit drugs.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2025-02-05 (Estimated); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
Number of sites with reduced probing depth | From the baseline (day 0) to post-treatment (day 45)
  Probing depth is determined as the distance from the gingival margin to the base of the pocket, measured at six sites per tooth: mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual, and disto-lingual.

SECONDARY OUTCOMES:
Number of sites with improved clinical attachment level | From the baseline (day 0) to post-treatment (day 45)
  The clinical attachment level is determined as the distance from the cementoenamel junction to the base of the pocket, measured at six sites per tooth: mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual, and disto-lingual.
Percentage of sites with bleeding on probing | From the baseline (day 0) to post-treatment (day 45)
  Bleeding on probing is evaluated 30 seconds after probing and recorded as present or absent at six sites per tooth: mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual, and disto-lingual.
Percentage of sites with biofilm | From the baseline (day 0) to post-treatment (day 45)
  The presence or absence of biofilm on the tooth surface, assessed at for sites per tooth (mesio, buccal, disto and lingual).
Number of teeth with dental mobility (by grade) | From the baseline (day 0) to post-treatment (day 45)
  Dental mobility is determined as the degree of movement of a tooth within its socket, assessed and recorded according to the following grades: Grade I (slight, up to 1 mm horizontal movement), Grade II (moderate, more than 1 mm horizontal movement), and Grade III (severe, includes vertical movement)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Franchin, PhD, Principal Investigator — Universidade Federal de Alfenas
Locations (1):
- Universidade Federal de Alfenas, Alfenas, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No